CLINICAL TRIAL: NCT02940691
Title: A Phase IV, Open-label, Single Arm, Multicentre Trial of Grazoprevir/Elbasvir for Genotype 1 or 4 in People With Chronic Hepatitis C Virus Infection and Recent Injecting Drug Use or Receiving Opioid Substitution Therapy
Brief Title: Scale-up of Treatment of Hepatitis C Infection Among People Who Inject Drugs
Acronym: DARLO-C
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor recruitment due to new treatments becoming available.
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1510
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Grazoprevir/elbasvir (Experimental): Grazoprevir/elbasvir (100mg/50mg) daily taken orally for 12 weeks.
  Interventions: Drug: Grazoprevir/elbasvir

INTERVENTIONS:
Drug: Grazoprevir/elbasvir — Grazoprevir/elbasvir (100mg/50mg) once daily for 12 weeks.
  Other Names: Zepatier

SUMMARY:
This study is a phase IV, open-label, single arm, multicentre study whose aim is to assess whether interferon-free and ribavirin-free Direct Acting Antiviral (DAA) Hepatitis C Virus (HCV) therapy with grazoprevir/elbasvir, will be feasible for the treatment of People who inject drugs (PWID) with recent injecting drug use or people receiving opioid substitution therapy and chronic HCV genotype 1 or 4 infection.

DETAILED DESCRIPTION:
A prospective, observational cohort design will be used to enrol patients attending tertiary, drug and alcohol and primary health care services in Sydney, Australia.

The study consists of a treatment phase (12 weeks) and a follow-up phase (up to 3 years) where participants will be followed every 3 months for the first year and every 6 months in years 2-3 to evaluate treatment response and reinfection.

The effectiveness of the treatment will be assessed by looking at the proportion of patients with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) following therapy with grazoprevir/elbasvir and evaluate demographic and clinical predictors of non-response.

ELIGIBILITY:
Inclusion Criteria:

* Participants have voluntarily signed the informed consent form.
* Be ≥18 years of age on day of signing informed consent form.
* Have chronic HCV genotype 1 or 4 infection (defined as detectable HCV RNA).
* Recent injecting drug use (previous 6 months) or receiving opioid substitution therapy.
* HIV-1 infected subjects enrolled in the study must meet the following criteria:

  * Have HIV infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry (Baseline) and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 p24 antigen, or plasma HIV-1 RNA viral load
  * b) Be on HIV Antiretroviral Therapy (ART) for at least 4 weeks prior to study entry using an ART regimen that is allowable with the intended DAA regimen as determined by the current PI and the Liverpool drug interaction website (http://www.hiv-druginteractions.org/) or current prescribing guidelines for elbasvir/grazoprevir OR be naive to treatment with any antiretroviral therapy (ART) with a baseline CD4 count of >200 and have no plans to initiate ART treatment while participating in this study and through to at least Follow-up Week 4.
* Negative pregnancy test at screening and baseline (females of childbearing potential only).
* All fertile males and females must be using effective contraception during treatment and during 14 days after treatment end.

Exclusion Criteria:

* Is taking or plans to take any prohibited medications as per DAA Product Information or herbal supplements, including but not limited to St. John's Wort (Hypericum perforatum) within 2 weeks of Baseline.
* Is currently using or intends to use barbiturates.
* Is a female and is pregnant or breast-feeding, or expecting to conceive or donate eggs from Baseline and continue throughout treatment, and after the last dose of study medication (as per the regimen requirements), or longer if dictated by local regulations.
* Has any condition or pre-study laboratory abnormality, ECG abnormality or history of any illness, which, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs to the subject.
* Had a life-threatening SAE during the screening period.
* Has exclusionary laboratory values as listed below:

  * Haemoglobin < 9.5 g/dL for both males and females
  * Platelets < 50 x 10^3 /µL
  * Serum albumin < 3.0 g/dL
* Patients with Child Pugh-B or C decompensated cirrhosis
* Previous HCV treatment-experience.
* Ongoing severe psychiatric disease as judged by the treating physician.
* Frequent injecting drug use that is judged by the treating physician to compromise treatment safety.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* Is Hepatitis B surface antigen (HBsAg) positive

NOTE: Sanger sequencing will be performed on a pre-treatment sample on all participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Dore, MBBS, Principal Investigator — Kirby Institute
Locations (5):
- Australia (5):
  - Kirketon Road Centre, Darlinghurst, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - The Langton Centre, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Drug and Alcohol Clinical Services (Hunter), Newcastle, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grebely J, Read P, Cunningham EB, Weltman M, Matthews GV, Dunlop A, Montebello M, Martinello M, Gilliver R, Marks P, Applegate TL, Dore GJ; DARLO-C Study Group. Elbasvir and grazoprevir for hepatitis C virus genotype 1 infection in people with recent injecting drug use (DARLO-C): An open-label, single-arm, phase 4, multicentre trial. Health Sci Rep. 2020 Mar 15;3(2):e151. doi: 10.1002/hsr2.151. eCollection 2020 Jun. PMID 32270056

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Grazoprevir/Elbasvir
Started | 32
Completed | 26
Not Completed | 6
Not completed — Lost to Follow-up | 5
Not completed — Incarceration | 1

BASELINE CHARACTERISTICS:
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  ≤46 years | 16
  >46 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 22
  Ethnicity: Non-caucasian | 10
Income [Count of Participants; unit: Participants]
  Full time employment | 0
  Part time employment | 1
  Disability/social services | 30
  Other | 1
Any non-injecting drug use in the previous month [Count of Participants; unit: Participants] | 11
Any injecting drug use in the previous month [Count of Participants; unit: Participants] | 29
Any alcohol use in the previous month [Count of Participants; unit: Participants] | 24
Hazardous alcohol use in the previous month [Count of Participants; unit: Participants] — Hazardous alcohol consumption is defined as a score of 3 or more for women and 4 or more for men on the Alcohol Use Disorders Identification Test (AUDIT-C).
  Participants | 23
History of opioid substitution therapy (OST) [Count of Participants; unit: Participants] | 23
Current opioid substitution therapy (OST) [Count of Participants; unit: Participants] | 18
Hepatitis C virus (HCV) genotype [Count of Participants; unit: Participants]
  1a | 29
  1b | 3
Stage of liver disease [Count of Participants; unit: Participants]
  No or mild fibrosis (F0-F1) | 23
  Moderate or advanced fibrosis (F2-F3) | 7
  Cirrhosis (F4) | 2

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HCV RNA at 12 Weeks Post End of Treatment (SVR12)
Description: Number with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) following 12 weeks of daily grazoprevir/elbasvir (100mg/50mg)
Time Frame: 12 weeks post treatment
Population: All enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 32
Participants
  SVR12 | 24
  No test performed | 2
  Lost to follow-up | 5
  Incarcerated | 1

2. Secondary Outcome: Number of Participants With Treatment Completion
Description: Number who completed HCV treatment as prescribed (12 weeks of grazoprevir/elbasvir (100mg/50mg) daily)
Time Frame: 12 weeks from treatment administration
Population: All enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 32
Participants
  Treatment completion | 26
  Lost to follow-up | 5
  Incarcerated | 1

3. Secondary Outcome: End of Treatment Response (Negative HCV RNA at the End of Treatment)
Description: Number with undetectable HCV RNA at end of treatment following 12 weeks of daily Grazoprevir/Elbasvir (100mg/50mg)
Time Frame: 12 weeks from treatment administration
Population: Those who completed treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir/Elbasvir
Number analyzed (Participants) | 26
Participants
  ETR | 24
  Not tested | 2

4. Other Pre Specified Outcome: Sensitivity and Specificity of the Finger-stick Xpert® HCV Viral Load Assay for HCV RNA Detection
Description: To determine the sensitivity and specificity of the Xpert® HCV Viral Load assay for HCV RNA detection in samples collected by finger-stick capillary whole-blood.
Time Frame: 12 week post treatment
Population: Only 22 had both Xpert and plasma samples collected. Some participants had >1 paired sample. HCV RNA from plasma was compared to the Xpert result. Sensitivity is number of positive Xpert results divided by the number of positive plasma results. The specificity is number of negative Xpert results divided by the number of negative plasma results.
Measure: Number (95% Confidence Interval); unit: Percentage
Units Other Than Participants: Samples
Groups:
- Xpert HCV VL Fingerstick: Sensitivity and specificity of the Xpert HCV VL Fingerstick assay for HCV detection in capillary whole-blood samples collected via fingerstick compares with Aptima HCV Quant Dx perforomed on EDTA plasma stored at -80C collected via venepuncture.
Arm/Group | Xpert HCV VL Fingerstick
Number analyzed (Participants) | 22
Number analyzed (Samples) | 36
Percentage
  Sensitivity | 100 [75.3 to 100]
  Specificity | 95.7 [78.1 to 99.9]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected in the study. Only serious adverse events were collected from Screening through to 4 weeks post end of treatment
Description: The studied medication was registered in the country of use and the study used the medication according to the indication. As the toxicity profile of this regimen is well known including within the patient population in this study, adverse events were not collected. Drug was accessed via the government subsidized medications program. Any adverse drug reactions were reported to the government health authority as per standard practice for medications supplied through the government program.
Arm/Group | Grazoprevir/Elbasvir
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir/Elbasvir (N=32)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Laceration of arm (Injury, poisoning and procedural complications) | 1 (1)
Schizoaffective Disorder (Psychiatric disorders) | 1 (1)
Drug-Induced Psychosis (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT02940691/Prot_SAP_000.pdf